CLINICAL TRIAL: NCT03640247
Title: Are Narcotic Pain Medications Necessary Following Thyroidectomy and Parathyroidectomy
Brief Title: Pain Medications Following Thyroidectomy and Parathyroidectomy
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: MetroHealth Medical Center (Other)
Responsible Party: Principal Investigator, Christopher McHenry, MD, Director, Division of General Surgery, MetroHealth Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-00412
Record Dates: First submitted 2018-07-24; First posted 2018-08-21 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Thyroid Disease; Parathyroid Diseases
Keywords: Thyroidectomy; Parathryoidectomy
MeSH Terms: conditions — Thyroid Diseases; Parathyroid Diseases | interventions — Ibuprofen; Acetaminophen; Oxycodone; Hydrocodone; Tramadol

STUDY DESIGN:
Masking Description: All party or parties involved have knowledge of the interventions assigned to individual participants
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Narcotic group regimen (Other): * Tylenol tablet 1000 mg by mouth every 8 hours alternating with
  * Ibuprofen tablet 800 mg by mouth every 8 hours
  * Oxycodone 5 mg by mouth every 6 hours as needed for pain, #10 tablet or if needed based on patient allergies, hydrocodone 5 mg/tramadol 50 mg.
  Interventions: Drug: Narcotic group regimen
- Non-narcotic group regimen (Active Comparator): * Tylenol tablet 1000 mg by mouth every 8 hours alternating with
  * Ibuprofen tablet 800 mg by mouth every 8 hours
  Interventions: Drug: Non-narcotic group regimen

INTERVENTIONS:
Drug: Non-narcotic group regimen — Non-Narcotic Group. Receives only alternating acetaminophen and ibuprofen
  Other Names: Ibuprofen 800mg every 8 hours; Acetaminophen 500Mg Tab x2 every 8 hours
  Arms: Non-narcotic group regimen
Drug: Narcotic group regimen — Narcotic Group: Alternating acetaminophen and ibuprofen, with a prescription of 10 tablets oxycodone (or if needed based on patient allergies, hydrocodone 5 mg/tramadol 50 mg) for break through pain.
  Other Names: Ibuprofen 800mg every 8 hours; Oxycodone 5mg every 6 hours prn for pain.; Hydrocodone 5 mg every 6 hours prn for pain; Tramadol 50 mg every 6 hours prn for pain; Acetaminophen 500Mg Tab x2 every 8 hours
  Arms: Narcotic group regimen

SUMMARY:
The purpose of this study is to evaluate the use of a non-narcotic, postoperative pain management regimen on patients undergoing thyroidectomy and parathyroidectomy.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the use of a non-narcotic, postoperative pain management regimen for patients undergoing thyroidectomy and parathyroidectomy. The investigators hypothesize that participants receiving non-narcotic pain regimens will have equivalent pain control and satisfaction to those who receive narcotic pain medicines.

The primary objective will be to identify if there is a difference in average perceived postoperative pain scores between participants who do and do not receive narcotic pain medications. Secondary outcomes will include need for breakthrough pain medications, patient satisfaction scores and the need to call the surgeon office for additional pain medications.

The participant will undergo total thyroidectomy, partial thyroidectomy or parathyroidectomy per the standard of care. The study will have no influence on the surgical procedure performed.

Following the surgery, postoperative analgesia regimens will be prescribed based on study randomization.

Narcotic group regimen (63 patients):

* Tylenol tablet 1000 mg by mouth every 8 hours alternating with
* Ibuprofen tablet 800 mg by mouth every 8 hours
* Oxycodone 5 mg by mouth every 6 hours as needed for pain, #10 tablets

Non-narcotic group regimen (63 patients):

* Tylenol tablet 1000 mg by mouth every 8 hours alternating with
* Ibuprofen tablet 800 mg by mouth every 8 hours

Participants will be asked to complete a survey each day for the initial 5 days postoperatively. Survey data includes:

* Average pain level using the 10-point visual analogue scale
* Ease of following the pain regimen using a 3-point liker scale
* Total dose of oral narcotics converted into oral morphine equivalents that were taken by participants post-operatively
* If the patient needed to call the office due to inadequately controlled pain

If the participants do not have adequate pain control with the non-narcotic regimen, they may be prescribed additional narcotic pain medication at the discretion of the PI and remain enrolled in the study.

The investigators will also review participants charts for information regarding any postoperative office calls regarding postoperative needs (i.e. for pain medications).

The medical surgical information below is gathered as standard of care for each surgical procedure and will also be collected as part of this procedure:

* Patient name, medical record number
* Patient demographics (age, gender, BMI, ASA score)
* Past medical History
* Past surgical history
* Past social history
* Preoperative medications (including steroids, anticoagulation, opioid use)
* Pre-operative diagnosis
* Procedure performed and pain medications administered in the post-ambulatory care unit
* Postoperative complications including need for readmission within 30 days
* Length of stay in hospital

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or greater
* Undergoing total thyroidectomy, partial thyroidectomy or parathyroidectomy at MetroHealth Medical Center

Exclusion Criteria:

* Patients taking narcotics prior to surgery
* Patients who are unable or unwilling to follow study protocol requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2018-11-15 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Overall mean pain as assessed by 10 point visual analogue scale from the 6 post operative day time points. | Overall mean pain score from 6 time points (Post operative days 0,1,2,3,4,5)
  10 point visual analogue scale- (0- no pain, 1-3 mild, 4-6 moderate pain, 7-10 severe pain).

SECONDARY OUTCOMES:
Patient satisfaction with the pain medication regimen as assessed by 3-point likert scale from the 6 post operative day time points. | Mean patient satisfaction score from 6 time points (Post operative days 0,1,2,3,4,5)
  3 point likert scale (1- easy to manage, 2- manageable but not easy 3- difficult to manage)
Total dose of oral narcotics converted into oral morphine equivalents (see below) that were taken by participants post-operatively | Mean oral morphine equivalents from 6 time points (Post operative days 0,1,2,3,4,5)
  Oral morphine equivalents(OMEQ):
  Hydrocodone 5mg =1 OMEQ
  Oxycodone 5mg = 1.5 OMEQ
  Hydromorphone 1mg = 4 OMEQ
  Codeine 5mg = 0.15 OMEQ
  Tramadol 5mg = 0.20 OMEQ
Mean number of office calls/contacts from the 6 post operative day time points. | Mean number of office calls/contacts from 6 time points (Post operative days 0,1,2,3,4,5)
  Mean number of office calls/contacts from participants from post operative day 0, 1,2,3,4,5.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher R McHenry, MD, Principal Investigator — MetroHealth Medical Center
Locations (1):
- MetroHealth Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Background] Fujii MH, Hodges AC, Russell RL, Roensch K, Beynnon B, Ahern TP, Holoch P, Moore JS, Ames SE, MacLean CD. Post-Discharge Opioid Prescribing and Use after Common Surgical Procedure. J Am Coll Surg. 2018 Jun;226(6):1004-1012. doi: 10.1016/j.jamcollsurg.2018.01.058. Epub 2018 Feb 28. PMID 29499361
- [Background] Hill MV, Stucke RS, Billmeier SE, Kelly JL, Barth RJ Jr. Guideline for Discharge Opioid Prescriptions after Inpatient General Surgical Procedures. J Am Coll Surg. 2018 Jun;226(6):996-1003. doi: 10.1016/j.jamcollsurg.2017.10.012. Epub 2017 Nov 30. PMID 29198638
- [Background] Long SM, Lumley CJ, Zeymo A, Davidson BJ. Prescription and Usage Pattern of Opioids after Thyroid and Parathyroid Surgery. Otolaryngol Head Neck Surg. 2019 Mar;160(3):388-393. doi: 10.1177/0194599818779776. Epub 2018 May 29. PMID 29807482
- [Background] Lou I, Chennell TB, Schaefer SC, Chen H, Sippel RS, Balentine C, Schneider DF, Moalem J. Optimizing Outpatient Pain Management After Thyroid and Parathyroid Surgery: A Two-Institution Experience. Ann Surg Oncol. 2017 Jul;24(7):1951-1957. doi: 10.1245/s10434-017-5781-y. Epub 2017 Feb 3. PMID 28160140
- [Background] Tan WH, Yu J, Feaman S, McAllister JM, Kahan LG, Quasebarth MA, Blatnik JA, Eagon JC, Awad MM, Brunt LM. Opioid Medication Use in the Surgical Patient: An Assessment of Prescribing Patterns and Use. J Am Coll Surg. 2018 Aug;227(2):203-211. doi: 10.1016/j.jamcollsurg.2018.04.032. Epub 2018 May 7. PMID 29746919
- [Derived] Brady JT, Dreimiller A, Miller-Spalding S, Gesang T, Sehgal AR, McHenry CR. Are narcotic pain medications necessary after discharge following thyroidectomy and parathyroidectomy? Surgery. 2021 Jan;169(1):202-208. doi: 10.1016/j.surg.2020.03.027. Epub 2020 May 14. PMID 32416981